CLINICAL TRIAL: NCT05996432
Title: Non-invasive, Image-Based, In-Vivo Assessment of Tumor Hypoxia to Guide Hypoxia-Driven Adaptive Radiation Therapy
Brief Title: Image-Based, In-Vivo Assessment of Tumor Hypoxia to Guide Hypoxia-Driven Adaptive Radiation Therapy
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Evan Osmundson, MD, PhD, Associate Professor of Radiation Oncology, Vanderbilt-Ingram Cancer Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: VICC-EDMDT23195
Record Dates: First submitted 2023-07-13; First posted 2023-08-18 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Brain Metastases
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Brain Neoplasms | interventions — Magnetic Resonance Spectroscopy; fluoromisonidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Locally Advanced Squamous Cell Carcinoma of the Head and Neck (Experimental): Participants will undergo magnetic resonance imaging (MRI) scans and positron emission tomography (PET) scans and administered the imaging agent 18F-fluoromisonidazole.
  Interventions: Procedure: Magnetic Resonance Imaging (MRI); Procedure: Positron Emission Tomography (PET); Drug: 18F-fluoromisonidazole
- Brain metastases (Experimental): Participants will undergo magnetic resonance imaging (MRI) scans and positron emission tomography (PET) scans and administered the imaging agent 18F-fluoromisonidazole.
  Interventions: Procedure: Magnetic Resonance Imaging (MRI); Procedure: Positron Emission Tomography (PET); Drug: 18F-fluoromisonidazole

INTERVENTIONS:
Procedure: Magnetic Resonance Imaging (MRI) — Participants will undergo Magnetic Resonance Imaging
Procedure: Positron Emission Tomography (PET) — Participants will undergo Positron Emission Tomography
Drug: 18F-fluoromisonidazole — Given by IV

SUMMARY:
This study will apply novel MRI approaches with established sensitivity to tissue oxygen consumption and perfusion to predict hypoxia-associated radiation resistance, manifested as tumor recurrence and progression post-treatment.

DETAILED DESCRIPTION:
Primary Objective:

- To validate non-invasive, MRI-based markers of tumor hypoxia in patients with brain metastases or head and neck cancer with and without evidence of tumor hypoxia identified by 18F-FMISO-PET-CT.

Secondary Objectives:

* To assess treatment-related changes in tumor and peritumoral tissue oxygen consumption and perfusion via non-invasive MRI.
* To evaluate the effect of pre-treatment and post-treatment (3 months) tumor hypoxia on tumor recurrence, progression, and radiation necrosis in patients with central nervous system metastases treated with standard of care stereotactic radiosurgery.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed head and neck squamous cell carcinoma or a clinical diagnosis of CNS-excluded nervous system neoplasm and disorder (brain metastases)
* Measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions, minimum size 7mm) with CT scan, MRI, or calipers by clinical exam
* ECOG performance status </=1 Karnofsky >/=70%
* Life expectancy of greater than 6 months
* The effects of 18F-FMISO on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and up until the day after 18F-FMISO administration. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception on the days of 18F-FMISO administration
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* History of allergic reactions attributed to compounds of similar chemical or biologic composition to 18F-FMISO
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Brain metastases >3.0 cm
* Dural-based metastases concerning for leptomeningeal disease
* Hemorrhage within the lesion of interest
* Patients presenting for radiation after surgical resection of brain metastasis/metastases or primary head and neck cancer (adjuvant radiotherapy)
* Prior or current known history of disease involving the brain other than brain metastases and including but not limited to; cerebrovascular disease (i.e., stroke or large vessel disease), brain hemorrhage (i.e., subarachnoid hemorrhage or intraparenchymal hemorrhage), Alzheimer's disease or dementia, Parkinson's disease, Multiple Sclerosis or schizophrenia
* Prior overlapping radiation fields
* Not suitable to undergo MRI because of; severe claustrophobia, presence of metallic objects or implanted medical devices in body (i.e., cardiac pacemaker, aneurysm clips, surgical clips, prostheses, artificial hearts, valves with steel parts, metal fragments, shrapnel, tattoos near the imaging site, or steel implants)
* Presence of any other co-existing condition which, in the judgment of the investigator, might increase the risk to the subject
* Presence of serious systemic illness, including uncontrolled intercurrent infection or psychiatric/social situations which may limit compliance with study requirements
* Not suitable to undergo MRI, including weight greater than 350lbs (common weight limit for the MRI table)
* Prisoners, children <18 years of age
* Prior overlapping radiation fields
* Not suitable to undergo MRI because of; severe claustrophobia, presence of metallic objects or implanted medical devices in body (i.e., cardiac pacemaker, aneurysm clips, surgical clips, prostheses, artificial hearts, valves with steel parts, metal fragments, shrapnel, tattoos near the imaging site, or steel implants)
* Presence of any other co-existing condition which, in the judgment of the investigator, might increase the risk to the subject
* Presence of serious systemic illness, including uncontrolled intercurrent infection or psychiatric/social situations which may limit compliance with study requirements
* Not suitable to undergo MRI, including weight greater than 350lbs (common weight limit for the MRI table)
* Prisoners, children <18 years of age
* The effects of 18F-FMISO on the developing infant are unknown. For this reason, nursing women will be excluded from the trial

Pregnant patients which will be identified as follows;

* Patients over the age of 60 do not require a pregnancy test per institutional guidelines. We anticipate this to be most of our patient population due to the age distribution of cancer patients.
* Patients under the age of 60 will be offered a point of care pregnancy test when seen in consult at the department of Radiation Oncology.
* Patients refusing pregnancy testing can sign a waiver stating that they refuse pregnancy testing but that they are not known to be pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-05-17 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Validate non-invasive, MRI-based markers of tumor hypoxia in patients with brain metastases or head and neck cancer with and without evidence of tumor hypoxia identified by 18F-FMISO-PET-CT | 1.5 years
  MRI assessed oxygen extraction fraction (OEF, %)

SECONDARY OUTCOMES:
Assess treatment-related changes in tumor and peritumoral tissue oxygen consumption and perfusion via non-invasive MRI | 4 years
  MRI assessed oxygen extraction fraction (OEF, %)

OTHER OUTCOMES:
Evaluate the effect of pre-treatment and post-treatment tumor hypoxia on outcome | 4 years
  Tumor recurrence
Evaluate the effect of pre-treatment and post-treatment tumor hypoxia on outcome | 4 years
  Radiation necrosis

CONTACTS AND LOCATIONS:
Overall Officials: Evan Osmundson, MD, PhD, Principal Investigator — Vanderbilt University/Ingram Cancer Center
Locations (1):
- Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Informed Consent Form (2024-02-18): https://cdn.clinicaltrials.gov/large-docs/32/NCT05996432/ICF_000.pdf